CLINICAL TRIAL: NCT01476917
Title: The ATLAST Long-Term Study. A Multicenter, Prospective, Long-Term Study of the Attune Sleep Apnea System for the Treatment of Obstructive Sleep Apnea (OSA)
Brief Title: The ATLAST Long-Term Study
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: ApniCure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11449
Record Dates: First submitted 2011-11-16; First posted 2011-11-22 (Estimated); Last update posted 2012-11-07 (Estimated); Status verified 2012-11

CONDITIONS: Obstructive Sleep Apnea (OSA)
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): Subjects that completed the ATLAST Study
  Interventions: Device: Attune Sleep Apnea System

INTERVENTIONS:
Device: Attune Sleep Apnea System — Observation of Attune Sleep Apnea System for use during sleep.

SUMMARY:
The Study is a multi-center, prospective, open label, single-arm, three-month, long-term study of the Attune Sleep Apnea System for the treatment of obstructive sleep apnea (OSA). The objective of the study is to monitor long-term use of the Attune Sleep Apnea System.

ELIGIBILITY:
Inclusion Criteria:

* Subject participated in the ATLAST Study, and completed the 28-day take-home period
* Subject understands the Study protocol and is willing and able to comply with Study requirements and sign the informed consent form.
* The study physician and investigator believe that study participation is appropriate for the subject.
* Subject has at least one molar in each of the four quadrants of the mouth (right upper, right lower, left upper, and left lower).

Exclusion Criteria:

* Female subjects who are pregnant or intend to become pregnant during the study period.
* Poor nasal patency as evidenced by the inability to breathe through the nose with the mouth closed.
* Oral cavity infection or any other oral or dental condition or problem that would limit subject use of the Attune Sleep Apnea System
* History of any OSA surgical treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2011-11; Primary Completion 2012-06 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Mean number of hours per night of device use over a 3-month period | Each night's use
  Nightly use will be monitored over a 3-month take-home period.

CONTACTS AND LOCATIONS:
Overall Officials: Ian Colrain, PhD, Principal Investigator — Stanford Research Institute (SRI)
Locations (6):
- United States (6):
  - REM Medical, Phoenix, Arizona
  - Penninsula Sleep Center (PSC), Burlingame, California
  - SRI International, Menlo Park, California
  - Sleep Disorders Center of Georgia, Atlanta, Georgia
  - SleepMed, Columbia, South Carolina
  - Sleep Medicine Associates of Texas (SMAT), Dallas, Texas